CLINICAL TRIAL: NCT05589389
Title: HS68-Meat and Pattern Study
Brief Title: Meat and Dietary Pattern Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Principal Investigator, David Baer, Supervisory Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HS68 - Meat And Pattern Study
Record Dates: First submitted 2022-10-11; First posted 2022-10-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to one or 24 possible treatment sequences.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High Healthy Eating Index Diet with Minimally Processed Meat (Experimental): Participants will consume a diet with a high Healthy Eating Index along with meat that is minimally processed.
  Interventions: Other: High Healthy Eating Index Diet with Minimally Processed Meat
- High Healthy Eating Index Diet with Further Processed Meat (Experimental): Participants will consume a diet with a high Healthy Eating Index along with meat that is further processed.
  Interventions: Other: High Healthy Eating Index Diet with Further Processed Meat
- Typical Healthy Eating Index Diet with Minimally Processed Meat (Experimental): Participants will consume a diet with a typical Healthy Eating Index along with meat that is minimally processed.
  Interventions: Other: Typical Healthy Eating Index Diet with Minimally Processed Meat
- Typical Healthy Eating Index Diet with Further Processed Meat (Experimental): Participants will consume a diet with a typical Healthy Eating Index along with meat that is further processed.
  Interventions: Other: Typical Healthy Eating Index Diet with Further Processed Meat

INTERVENTIONS:
Other: High Healthy Eating Index Diet with Minimally Processed Meat — Participants will consume a diet with a high Healthy Eating Index along with meat that is minimally processed.
  Arms: High Healthy Eating Index Diet with Minimally Processed Meat
Other: High Healthy Eating Index Diet with Further Processed Meat — Participants will consume a diet with a high Healthy Eating Index along with meat that is further processed.
  Arms: High Healthy Eating Index Diet with Further Processed Meat
Other: Typical Healthy Eating Index Diet with Minimally Processed Meat — Participants will consume a diet with a typical Healthy Eating Index along with meat that is minimally processed.
  Arms: Typical Healthy Eating Index Diet with Minimally Processed Meat
Other: Typical Healthy Eating Index Diet with Further Processed Meat — Participants will consume a diet with a typical Healthy Eating Index along with meat that is further processed.
  Arms: Typical Healthy Eating Index Diet with Further Processed Meat

SUMMARY:
The objective of this study is to investigate how different types of meat consumed with two different dietary patterns affect risk for disease.

DETAILED DESCRIPTION:
Association studies have suggested that dietary meat intake may have negative impacts on health. However, these association studies have done a poor job separating meat intake from overall dietary pattern, as well as isolating effects of processed meat from minimally processed meat. Meat is a good source of several essential nutrients, including high quality protein, iron, and vitamin B12. This dietary intervention is designed to investigate the effects of minimally processed meat and further proceeded meat, as part of two different dietary patterns (the typical American dietary pattern and Dietary Guidelines dietary pattern) on outcomes related to chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female

Exclusion Criteria:

* Younger than 25 years old and older than 80 years old at the beginning of the intervention.
* Body mass index less than 18 or greater than 40 kg/m2.
* Blood pressure greater than 160/100 mm Hg or use of medication to treat hypertension for less than 6 months.
* Use of medications that will affect the study outcomes, including cholesterol lowering medications.
* Pregnant women, lactating women, women who plan to become pregnant during the study, or women who have given birth during the previous 12 months.
* Fasting blood glucose over 125 mg/dL or type 2 diabetes requiring medication.
* Body weight change of 10% in the past 3 months.
* History of bariatric or other gastrointestinal surgery that would affect digestion.
* History or presence of diabetes, kidney disease, liver disease, certain cancers, gout, hyperthyroidism, untreated or unstable hypothyroidism, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes.
* Smokers, vapers, or other tobacco users (within 6 months prior to the start of the study).
* Use of an antibiotic within 1 month of the start of the study or during the study.
* Plans to have a colonoscopy during the study.
* Allergy to any food included in the study menus.
* Unable or unwilling to give informed consent or communicate with study staff.
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion).
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Carnitine Concentration | Day 1
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 2
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 35
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 36
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 70
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 71
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 105
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 106
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 140
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Carnitine Concentration | Day 141
  Carnitine, which plays a role to reduce oxidative stress, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 1
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 2
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 35
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 36
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 70
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 71
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 105
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 106
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 140
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Choline Concentration | Day 141
  Choline, a molecule involved in methyl transfer and lipid formation and support of healthy blood vessels, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 1
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 2
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 35
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 36
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 70
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 71
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 105
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 106
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 140
  Betaine, which helps make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Betaine Concentration | Day 141
  Betaine, which help make carnitine and supports heart health, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 1
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 2
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 35
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 36
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 70
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 71
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 105
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 106
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 140
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMA (trimethylamine) Concentration | Day 141
  TMA (trimethylamine), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 1
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 2
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 35
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 36
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 70
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 71
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 105
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 106
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 140
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
TMAO (trimethylamine N-oxide) Concentration | Day 141
  TMAO (trimethylamine N-oxide), a metabolite of gastrointestinal bacteria, will be analyzed in blood in units of micromol/L to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 1
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 2
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 35
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 36
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 70
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 71
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 105
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 106
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 140
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Total Cholesterol Concentration | Day 141
  Total cholesterol will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 1
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 2
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 35
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 36
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 70
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 71
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 105
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 106
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 140
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
LDL Cholesterol Concentration | Day 141
  LDL cholesterol, including its subfractions LDL1, LDL2, LDL3, and LDL4, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 1
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 2
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 35
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 36
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 70
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 71
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 105
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 106
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 140
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
HDL Cholesterol Concentration | Day 141
  HDL cholesterol, including its subfractions HDL2 and HDL3, will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 1
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 2
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 35
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 36
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 70
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 71
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 105
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 106
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 140
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Triglyceride Concentration | Day 141
  Triglycerides will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 1
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 2
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 35
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 36
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 70
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 71
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 105
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 106
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 140
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Apolipoprotein Concentration | Day 141
  Apolipoproteins AI, AII, and B will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 1
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 2
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 35
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 36
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 70
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 71
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 105
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 106
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 140
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Lipoprotein(a) (Lp(a)) Concentration | Day 141
  Lipoprotein(a) will be analyzed in blood in units of mg/dl to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 1
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 2
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 35
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 36
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 70
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 71
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 105
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 106
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 140
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Low Density Lipoprotein particle size | Day 141
  Low Density Lipoprotein particle size will be analyzed in blood in units of nm to assess the effect of the intervention on cardiovascular health.
Blood Pressure | Day 1
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 2
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 35
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 36
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 70
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 71
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 105
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 106
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 140
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.
Blood Pressure | Day 141
  Blood pressure (systolic and diastolic) will be measured as mm Hg, as a reflection of cardiovascular health.

SECONDARY OUTCOMES:
Gut microbiota | Day 1
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 2
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 35
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 36
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 70
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 71
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 105
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 106
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 140
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Gut microbiota | Day 141
  Fecal samples will be analyzed for bacterial RNA sequences. Bacterial RNA sequences will reflect those bacteria (gut microbiota) who are actively expressing genes (and data will be expressed as operational taxonomic units) and will also reflect which genes are actively being expressed (and data will be expressed as RNA sequences).
Bile acid Concentration | Day 1
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 2
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 35
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 36
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 70
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 71
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 105
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 106
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 140
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Bile acid Concentration | Day 141
  Fecal samples will be analyzed for bile acids (cholic acid, chenodeoxycholic acids, lithocholic acid, and deoxycholic acids) and will be expressed in micromoles. Bile acids reflect gut bacterial activity and impact cancer and other health conditions.
Glucose Concentration | Day 1
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 2
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 35
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 36
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 70
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 71
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 105
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 106
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 140
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Glucose Concentration | Day 141
  Glucose in blood will be measured in mg/dL as a reflection of glucose regulation.
Insulin Concentration | Day 1
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 2
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 35
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 36
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 70
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 71
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 105
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 106
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 140
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Insulin Concentration | Day 141
  Insulin will be measured in blood in units of microIU/ml as a reflection of glucose regulation.
Diet Satisfaction | Week 1
  Diet satisfaction will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters, with higher values representing higher satisfaction.
Diet Satisfaction | Week 4
  Diet satisfaction will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters, with higher values representing higher satisfaction.
Diet Satisfaction | Week 5
  Diet satisfaction will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters, with higher values representing higher satisfaction.
Diet Satisfaction | Week 9
  Diet satisfaction will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters, with higher values representing higher satisfaction.
Diet Satisfaction | Week 10
  Diet satisfaction will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters, with higher values representing higher satisfaction.
Diet Satisfaction | Week 14
  Diet satisfaction will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters, with higher values representing higher satisfaction.
Diet Satisfaction | Week 15
  Diet satisfaction will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters, with higher values representing higher satisfaction.
Diet Satisfaction | Week 19
  Diet satisfaction will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters, with higher values representing higher satisfaction.
Hunger and Satiety | Week 1
  Hunger and satiety will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters. Higher mm values for hunger indicate greater hunger; higher mm values for satiety indicate greater satiety.
Hunger and Satiety | Week 4
  Hunger and satiety will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters. Higher mm values for hunger indicate greater hunger; higher mm values for satiety indicate greater satiety.
Hunger and Satiety | Week 5
  Hunger and satiety will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters. Higher mm values for hunger indicate greater hunger; higher mm values for satiety indicate greater satiety.
Hunger and Satiety | Week 9
  Hunger and satiety will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters. Higher mm values for hunger indicate greater hunger; higher mm values for satiety indicate greater satiety.
Hunger and Satiety | Week 10
  Hunger and satiety will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters. Higher mm values for hunger indicate greater hunger; higher mm values for satiety indicate greater satiety.
Hunger and Satiety | Week 14
  Hunger and satiety will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters. Higher mm values for hunger indicate greater hunger; higher mm values for satiety indicate greater satiety.
Hunger and Satiety | Week 15
  Hunger and satiety will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters. Higher mm values for hunger indicate greater hunger; higher mm values for satiety indicate greater satiety.
Hunger and Satiety | Week 19
  Hunger and satiety will be measured by questionnaire using a visual analogue scale, with responses measured in millimeters. Higher mm values for hunger indicate greater hunger; higher mm values for satiety indicate greater satiety.
24-Hour Dietary Recall | 5 to 7 days before Day 1
  Prior to the start of the intervention, a 24-hour dietary recall interview will be conducted to assess food intake during the previous day. Data will be expressed as specific foods and how much of each food (grams) was consumed. The assessment will occur prior to the start of the dietary intervention, during baseline measurements, at approximately 5 to 7 days, and at approximately 3 to 5 days, and at approximately 1 to 3 days before the start of the dietary intervention (week 1).
24-Hour Dietary Recall | 3 to 5 days before Day 1
  Prior to the start of the intervention, a 24-hour dietary recall interview will be conducted to assess food intake during the previous day. Data will be expressed as specific foods and how much of each food (grams) was consumed. The assessment will occur prior to the start of the dietary intervention, during baseline measurements, at approximately 5 to 7 days, and at approximately 3 to 5 days, and at approximately 1 to 3 days before the start of the dietary intervention (week 1).
24-Hour Dietary Recall | 1 to 3 days before Day 1
  Prior to the start of the intervention, a 24-hour dietary recall interview will be conducted to assess food intake during the previous day. Data will be expressed as specific foods and how much of each food (grams) was consumed. The assessment will occur prior to the start of the dietary intervention, during baseline measurements, at approximately 5 to 7 days, and at approximately 3 to 5 days, and at approximately 1 to 3 days before the start of the dietary intervention (week 1).
IL6 Concentration | Day 1
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 2
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 35
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 36
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 70
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 71
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 105
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 106
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 140
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
IL6 Concentration | Day 141
  IL6, which is a measure of inflammation, will be measured in blood in units of pg/ml.
C-Reactive Protein (CRP) Concentration | Day 1
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 2
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 35
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 36
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 70
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 71
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 105
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 106
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 140
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
C-Reactive Protein (CRP) Concentration | Day 141
  C-Reactive Protein, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 1
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 2
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 35
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 36
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 70
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 71
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 105
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 106
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 140
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.
Serum Amyloid A Concentration | Day 141
  Serum Amyloid A, which is a measure of inflammation, will be measured in blood in units of ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: David J. Baer, PhD, Principal Investigator — USDA Beltsville Human Nutrition Research Center; Janet A. Novotny, PhD, Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No